CLINICAL TRIAL: NCT02232984
Title: Quadripolar CRT-D On Currently Approved Lead SystemS
Acronym: CROSS X4
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CROSSX4
Record Dates: First submitted 2014-08-27; First posted 2014-09-08 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiac Resynchronization Therapy (CRT); CRT-D; Quadripolar pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All study patients: All study patients will be implanted with a Boston Scientific (BSC) quadripolar Cardiac Resynchronization Therapy (CRT-D) and a currently approved quadripolar left ventricular lead. At the pre-discharge visit, multiple vectors will be tested in order to assess their respective performance.

SUMMARY:
The purpose of the study is to evaluate different ways to program around extracardiac stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is medically indicated for implantation with a Boston Scientific (BSC) DYNAGEN or INOGEN X4 CRT-D (or any future FDA approved BSC X4 CRT-D) and already implanted with/scheduled to receive a commercially available quadripolar left ventricular lead
* Subject is willing and capable of providing informed consent and participating in all testing and study visits associated with this investigation at an approved center and at the intervals defined by this protocol
* Subject is age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Subject has a known or suspected sensitivity to dexamethasone acetate (DXA)
* Subject is enrolled in any other concurrent study, without prior approval from BSC
* Women of childbearing potential who are or might be pregnant at the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from the center's general population who are indicated for a CRT-D. All study subjects will be implanted with the BSC DYNAGEN or INOGEN X4 CRT-D (or any future FDA approved BSC X4 CRT-D). Subjects may have a previously implanted/will be receiving an approved quadripolar left ventricular lead.
Sampling Method: Probability Sample
Enrollment: 749 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Ellis, MD, Principal Investigator — Vanderbilt University Medical Center, Nashville, TN
Locations (60):
- United States (60):
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Phoenix Cardiovascular Research Group/ Heart & Vascular Center of Arizona, Phoenix, Arizona
  - St. Joseph's Hospital, Phoenix, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - Cardiology Associates of Northeast Arkansas, Jonesboro, Arkansas
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Comprehensive Cardiovascular Medical Group, Bakersfield, California
  - Cardiac Device Rhythm Specialists, Inc, Los Angeles, California
  - Desert Heart Rhythm, Palm Springs, California
  - Bradenton Cardiology Center, Bradenton, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - North Florida VA, Gainesville, Florida
  - Northeast Cardiology Clinic, Jacksonville, Florida
  - Watson Center Clinic for Research, Lakeland, Florida
  - Charlotte Heart, Port Charlotte, Florida
  - Brevard Cardiovascular Res. Associates, Rockledge, Florida
  - Central Florida Regional, Sanford, Florida
  - Sarasota Memorial Hosptial, Sarasota, Florida
  - Northside Hospital, St. Petersburg, Florida
  - Tallahassee Memorial, Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta Heart Specialist, Atlanta, Georgia
  - AnMed Health, Augusta, Georgia
  - University Hospital, Augusta, Georgia
  - North Georgia Heart Foundation, Gainesville, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - West Suburban Hospital, Oak Park, Illinois
  - Central DuPage Medical Center, Winfield, Illinois
  - Lutheran Hospital, Fort Wayne, Indiana
  - Parkview Hospital, Fort Wayne, Indiana
  - Community Hospital, Munster, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Ark-La-Tex Cardiology, APMC, Shreveport, Louisiana
  - Willis Knighton, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Hospital, Flint, Michigan
  - Genesys Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Lakeland Medical Center, Saint Joseph, Michigan
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - Desert Springs, Las Vegas, Nevada
  - Catholic Medical Center, Manchester, New Hampshire
  - Atlanticare Regional Medical Center, Atlantic City, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mercy Hospital/ Buffalo Heart Group, Buffalo, New York
  - Genesis Health System, Zanesville, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Mercer Bucks Cardiology, Newtown, Pennsylvania
  - Regional Hospital of Scranton, Scranton, Pennsylvania
  - Core CV Research, Jackson, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Arrhythmia Associates, Houston, Texas
  - Houston Cardiovascular Associates, Houston, Texas
  - Heart Institute of East Texas, Lufkin, Texas
  - Woodlands North Houston Heart Ctr, The Woodlands, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Hunter Holmes VA Medical Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Belin Healthcare, Green Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 749 subjects were enrolled. Of these, 7 did not complete baseline demographics due to early withdrawals and 1 additional was withdrawn due to LV lead not placed. Therefore, baseline demographics is based on a maximum of 742 subjects.
Groups:
- All Study Patients: All study patients were implanted with a BSC quadripolar CRT-D and a currently approved quadripolar left ventricular lead. At the pre-discharge visit, multiple vectors were tested in order to assess their respective performance.
Period: Overall Study
Arm/Group | All Study Patients
Started | 749 (Enrolled subjects)
Successfully Implanted | 675 (Successfully implanted subjects)
Completed | 672 (Total number of subjects who completed study)
Not Completed | 77
Not completed — Withdrawal by Subject | 5
Not completed — Death | 1
Not completed — Investigator withdrawal | 10
Not completed — Device implant unsuccessful | 53
Not completed — not disclosed by site | 7
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Of the 749 enrolled subjects, 742 subjects provided baseline demographics information. Six were early withdrawals and one additional was not implanted with LV lead.
Arm/Group | All Study Patients
Number analyzed (Participants) | 742
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180
  Male | 562
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 742
Left Ventricular Ejection Fraction (LVEF) % [Mean (Standard Deviation); unit: %] — Population: Number of subjects with this baseline characteristic is smaller than overall population because this information was not collected/provided by the centers for all patients.
  %
    number analyzed (Participants) | 738
    (all) | 26.5 (8.3)
QRS width [Mean (Standard Deviation); unit: ms] — Population: Number of subjects with this baseline characteristic is smaller than overall population because this information was not collected/provided by the centers for all patients.
  ms
    number analyzed (Participants) | 736
    (all) | 153.7 (28.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Vectors With Phrenic Nerve Stimulation (PNS)
Description: The primary objective of this study was to characterize the performance of Boston Scientific (BSC) unique pacing vectors vs. BSC/St Jude Medical (STJ) common pacing vectors to prevent phrenic nerve stimulation (PNS) based on the selected pacing cathode. BSC unique vectors are those that are only available with Boston Scientific's (BSC) quadripolar (X4) CRT-Ds while common vectors are those that are available for both BSC and STJ systems.
Time Frame: Pre-discharge (up to 7 days post implant)
Measure: Number; unit: Number of Pacing vectors with PNS
Arm/Group | All Study Patients
Number analyzed (Participants) | 672
Number of Pacing vectors with PNS
  Unique pacing vectors with PNS | 181
  Common vectors with PNS | 189

2. Secondary Outcome: Final Pacing Treshold at Pre-discharge
Description: Characterize the electrical performance of BSC pacing vectors using pacing thresholds. Summary statistics for LV Tip1 to LV Ring 2 pacing thresholds for the BSC pacing vectors were reported. The electrical measurements were taken using the implanted pulse generator (PG) per standard practice.
Time Frame: Pre-discharge (up to 7 days post implant)
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | All Study Patients
Number analyzed (Participants) | 672
Volts | 1.93 (1.87)

3. Secondary Outcome: Final LV Lead Impedance at Pre-discharge
Description: Characterize the electrical performance of BSC pacing vectors using impedance measurements. Summary Statistics Were Provided for LV Tip 1 to LV Ring 2 Measurements. The electrical measurements were taken using the implanted pulse generator (PG) per standard practice.
Time Frame: Pre-discharge (up to 7 days post implant)
Measure: Mean (Standard Deviation); unit: Ohms
Groups:
- All Study Patients: All study patients were implanted with a BSC quadripolar CRT-D and a currently approved quadripolar left ventricular lead. At the pre-discharge visit, multiple vectors were be tested in order to assess their respective performance. Performance of the LV lead delivery system (Acuity Pro vs other LV delivery systems) were assessed. Although use of Acuity Pro was recommended, choice of delivery system was at the physician's discretion.
Arm/Group | All Study Patients
Number analyzed (Participants) | 672
Ohms | 1034.7 (310.6)

4. Secondary Outcome: Final Sensing Amplitude at Pre-discharge
Description: Characterize the electrical performance of BSC pacing vectors using sensing amplitudes. Summary statistics were provided for LV Tip 1 to LV Ring 2 measurements. The electrical measurements were taken using the implanted pulse generator (PG) per standard practice.
Time Frame: Pre-discharge (up to 7 days post implant)
Measure: Mean (Standard Deviation); unit: Milivolts
Arm/Group | All Study Patients
Number analyzed (Participants) | 672
Milivolts | 13.30 (6.40)

5. Secondary Outcome: Delivery System Comparison Between ACUITY Pro and the Other Delivery Systems
Description: Characterize the performance of the BSC ACUITY Pro delivery system versus competitive delivery systems in the placement of LV leads. Data collected on the use of the ACUITY Pro delivery system and competitive systems were characterized by presenting summary statistics by system (all competitive devices maybe combined for purposes of reporting), and differences between the ACUITY Pro system and competitive systems were reported as appropriate.
Time Frame: At time of implantation (0 to 30 days post consent signature)
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Acuity Pro LV Lead Delivery System: All study patients were implanted with a BSC quadripolar CRT-D and a currently approved quadripolar left ventricular lead. At the pre-discharge visit, multiple vectors were be tested in order to assess their respective performance. Performance of the LV lead delivery system (Acuity Pro vs other LV delivery systems) were assessed. Although use of Acuity Pro was recommended, choice of delivery system was at the physician's discretion.
- Other LV Lead Delivery Systems: All study patients were implanted with a BSC quadripolar CRT-D and a currently approved quadripolar left ventricular lead. At the pre-discharge visit, multiple vectors will be tested in order to assess their respective performance. Performance of the LV lead delivery system (Acuity Pro vs other LV delivery systems) was assessed. Although use of Acuity Pro was recommended, choice of delivery system was at the physician's discretion.
Arm/Group | Acuity Pro LV Lead Delivery System | Other LV Lead Delivery Systems
Number analyzed (Participants) | 394 | 281
Minutes
  Skin to skin time (min) | 82.4 (38.9) | 87.8 (38.9)
  Lead placement time (min) | 24.5 (23.5) | 29.8 (24.8)
  CS Canulation Time (min) | 6.2 (9.4) | 7.8 (12.2)
  Overall catheter in the body time (min) | 25.9 (21.8) | 32.7 (25.1)

ADVERSE EVENTS:
Time Frame: From enrollment through pre-discharge (up to 7 days post-implant). Study was completed at pre-discharge.
Groups:
- All Study Patients: All study patients were implanted with a BSC quadripolar CRT-D and a currently approved quadripolar left ventricular lead. At the pre-discharge visit, multiple vectors were be tested in order to assess their respective performance.
Arm/Group | All Study Patients
All-Cause Mortality (participants affected / at risk) | 1/749
Serious Adverse Events (participants affected / at risk) | 16/749
Other Adverse Events (participants affected / at risk) | 11/749
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Patients (N=749)
Adverse reaction - general (Injury, poisoning and procedural complications) | 1 (1)
Adverse drug reaction - respiratory (Injury, poisoning and procedural complications) | 1 (1)
Inadvertent VT/VF (Cardiac disorders) | 2 (2)
Hematoma pocket <= 30 days (Injury, poisoning and procedural complications) | 1 (1)
Dislodgement - undersensing RV (Cardiac disorders) | 1 (1)
Dislodgement - no reported signs - RA (Cardiac disorders) | 4 (4)
Elevated threshold - RV (Cardiac disorders) | 1 (1)
Dislodgment - no reported signs - LV (Cardiac disorders) | 3 (3)
Coronary venous dissection (Injury, poisoning and procedural complications) | 1 (1)
Dislodgment - no reported signs - RV (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Patients (N=749)
Dislodgement - no reported signs - RA (Cardiac disorders) | 5 (5)
Coronary Venous dissection (Injury, poisoning and procedural complications) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No